CLINICAL TRIAL: NCT02857387
Title: Markers of Vascular Aging and Coronary Syndrome
Acronym: MAVASCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PO15043
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

ARMS (1):
- acute coronary syndrome (Experimental)
  Interventions: Biological: blood sample withdrawn

INTERVENTIONS:
Biological: blood sample withdrawn

SUMMARY:
Atherosclerosis and aging are associated to the raise of biochemical alterations of proteins grouped under the name of " non-enzymatic post-translational modifications ". They often correspond to the irreversible binding of glucose or other oses (glycation) or urea derivatives (carbamylation) on proteins and lead to the formation of complex compounds (post-translational modifications derived products, PTMD) that can accumulate in tissues and be responsible for deleterious effects. The specific role of these compounds in the pathophysiology of aging and atherosclerosis remains unknown, as are the molecular and cellular mechanisms implicated.

This project is based on the hypothesis that non-enzymatic post-translational modifications may cause changes in the genesis of complication of coronary atherosclerosis and that PTMD could therefore constitute relevant biomarkers in this specific clinical situation.

To explore these potential new biomarkers, the investigators designed a study in patients having experienced an acute coronary syndrome and followed during a year. The concentrations of PTMD assayed at 0, 1, 3, 12 months, will be correlated to clinical (severity and evolution) and paraclinical (cutaneous autofluorescence) data and the effect of cardiac rehabilitation will be assessed.

This should help to identify new (and non-traditional) biomarkers of coronary heart disease and determine some of the implicated pathophysiological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary heart syndrome
* included during hospitalization, usual cardiologic follow-up planned in Reims university hospital

Exclusion Criteria:

* <18yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Post-translational modifications of Proteins quantification assessed by Liquid chromatography-mass spectrometry | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France